CLINICAL TRIAL: NCT07351344
Title: African Survey on Sepsis Knowledge (ASK)
Acronym: ASK
Status: Recruiting | Type: Observational
Sponsor: Claudia Spies (Other)
Responsible Party: Sponsor-Investigator, Claudia Spies, Head of the Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charité - University Medicine Berlin, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: STAIRS
Record Dates: First submitted 2025-12-16; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants from the first wave: 150 adult participants from healthcare professions from partner institutions in Uganda, Ethiopia, the Democratic Republic of Congo, Mozambique, Ghana, Sierra Leone, and Nigeria are surveyed.
- Participants from the second wave: 150 adult participants from healthcare professions from partner institutions in Uganda, Ethiopia, the Democratic Republic of Congo, Mozambique, Ghana, Sierra Leone, and Nigeria are surveyed.

SUMMARY:
This study is an anonymous online survey on clinical knowledge of sepsis among healthcare professionals in seven countries in sub-Saharan Africa. The survey is to be repeated every 12-24 months.

DETAILED DESCRIPTION:
The survey is being conducted in the partner countries of the research network "sub-Saharan Africa consorTium for the Advancement of Innovative Research and Care in Sepsis (STAIRS)," which is funded by the German Federal Ministry of Research, Technology and Space (BMFTR). As part of clinical capacity building in partner institutions in Uganda, Ethiopia, the Democratic Republic of the Congo, Mozambique, Ghana, Sierra Leone, and Nigeria, the project will establish a series of webinars and a learning platform, among other things. The survey will be conducted in two separate cross-sectional waves. The baseline survey serves to identify relevant knowledge gaps and determine the needs of various groups of healthcare professionals. The second wave will compare sepsis knowledge scores between waves.

ELIGIBILITY:
Inclusion Criteria:

* Occupation: adult members of a healthcare profession (e.g., doctors, nurses, midwifes) or their trainees
* Place of work: employment in a healthcare facility in one of the seven partner countries (Uganda, Ethiopia, Democratic Republic of the Congo, Mozambique, Ghana, Sierra Leone, Nigeria).
* Consent: Willingness to participate voluntarily in the anonymous online survey.

Exclusion Criteria:

* Not employed in a healthcare profession (e.g., administrative staff, non-medical professionals)
* Not employed in one of the participating countries. Incomplete questionnaires (< 50% of questions answered)
* No internet access or technical limitations that make participation impossible. To complete the survey online.
* Language skills: Sufficient language skills in the survey language (English or French)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult members of a healthcare profession (e.g., doctors, nurses, clinical officers) or their trainees from healthcare facility in one of the seven partner countries (Uganda, Ethiopia, Democratic Republic of the Congo, Mozambique, Ghana, Sierra Leone, Nigeria).
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Sepsis - Knowledge - Score | Baseline survey period (January 19, 2026 - April 30, 2026) and follow-up survey period (April 1, 2027 - July 31, 2027)
  * Measured as the sum of correctly answered questions in the questionnaire. This results in a sepsis knowledge score of 0-47 points, with higher scores indicating better knowledge.
  * Assessed in two independent cross-sectional survey waves.
  * Calculated for all participants.
  * Serves as the main measure of clinical sepsis knowledge in partner countries across survey waves conducted before and after the implementation period of capacity-building activities

SECONDARY OUTCOMES:
Domain-specific knowledge of sepsis | Baseline survey period (January 19, 2026 - April 30, 2026), and follow-up survey period (April 1, 2027 - July 31, 2027)
  Domain-specific knowledge of sepsis is measured in five domains, to identify specific knowledge gaps. Domain-specific scores will be measured as the sum of correctly answered questions in the questionnaire in respective domain. Domains are:
  1. definitions of sepsis and septic shock (0-8 points, with higher points indicating higher knowledge)
  2. sepsis risk groups (0-6 points, with higher points indicating higher knowledge),
  3. causes of sepsis (0-6 points, with higher points indicating higher knowledge),
  4. sepsis symptoms (0-6 points, with higher points indicating higher knowledge),
  5. management of sepsis (0-21 points, with higher points indicating higher knowledge).
  All domains together sum up to the overall sepsis knowledge score (primary outcome).
Analysis of sepsis knowledge scores and domain-specific scores by professional role | Baseline survey period (January 19, 2026 - April 30, 2026), and follow-up survey period (April 1, 2027 - July 31, 2027)
  * Correlations between sepsis knowledge scores and professional roles and different levels of education within professional groups (nurses, doctors, and midwifes).
  * Regression-based predictors of overall sepsis knowledge scores and domain-specific scores by professional roles and different levels of education within the professional groups of nurses, doctors, and midwifes
Country comparison | Baseline survey period (January 19, 2026 - April 30, 2026), and follow-up survey period (April 1, 2027 - July 31, 2027)
  • Between group comparison in sepsis knowledge scores and domain-specific sepsis knowledge between different countries (Uganda, Ethiopia, the Demoratic Republic of the Congo, Mozambique, Ghana, Sierra Leone, Nigeria, (potentially other countries in case of spill-over).
Second survey wave only: Change in sepsis knowledge scores between survey waves | Follow-up survey period (April 1, 2027 - July 31, 2027)
  - Difference in average knowledge score in repeated survey.
  * Between-wave comparison of sepsis knowledge scores and domain specific sepsis knowledge scores in a comparison between baseline assessment and after implementation of STAIRS capacity building measures
  * Comparisons between survey waves will be conducted using appropriate parametric or non-parametric tests
Comparison of sepsis knowledge scores by self-reported participation in capacity-building measures | Follow-up survey period (April 1, 2027 - July 31, 2027)
  * Comparison of sepsis knowledge scores and domain-specific scores between respondents who report participation in capacity-building activities and those who do not
  * If possible, assessment of correlations and adjusted relationships between participation in capacity-building activities and sepsis knowledge scores
Baseline survey only: Self-assessment of perceived training needs | Baseline survey period (January 19, 2026 - April 30, 2026)
  * Exploratory analysis of self-reported sepsis training needs, and preferred formats (virtual vs. in-person)
  * Self-reported perception of the importance of sepsis as a training subject
Vignette-based sepsis knowledge score (sum of correct responses to predefined vignette items) | Baseline survey period (January 19, 2026 - April 30, 2026), and follow-up survey period (April 1, 2027 - July 31, 2027)
  * Calculated as the sum of correct responses (0-9 points) to predefined items across four clinical case vignettes
  * Analyzed separately from the primary sepsis knowledge score
  * Analyzed descriptively and compared between groups and survey waves using appropriate statistical tests

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charité - University Medicine Berlin
Locations (1):
- The Komfo Anokye teaching hospital, Kumasi, Ghana

IPD SHARING:
Plan to Share IPD: No